CLINICAL TRIAL: NCT06367959
Title: Health Benefits of Writing Therapy Among Asian American Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0324; NCI-2024-02939 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control condition (Experimental): Participants will be asked to write about facts regarding their cancer diagnosis and treatment in writing sessions.
  Interventions: Behavioral: Esays; Behavioral: Questionnaires
- Intervention Condition (Experimental): Participants will be asked to write about different topics regarding their cancer experience. During session 1, participants will be asked to write about the stress of having cancer and their strategies for coping with stressors associated with their cancer (i.e., stress and coping). During session 2, participants will be asked to write about their deepest feelings regarding their cancer experience (i.e., emotional disclosure). During session 3 and the booster session (at 9-month follow-up), participants will be asked to write about positive thoughts and feelings regarding their experience with cancer.
  Interventions: Behavioral: Esays; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Esays — Participants will write about their experiences One (1) time each week for 3 weeks at the beginning of the study and then 1 more time 9 months later. Participants will be asked to write about their experiences with cancer in English or Chinese and to write as much as they can for about 20-30 minutes for each essay.
Behavioral: Questionnaires — Participants will answer a questionnaire at the beginning of the study and then 3, 6, and 12 months later.
  Participants will also answer a questionnaire about their thoughts on writing and on the study after they complete the third essay.

SUMMARY:
To learn more about participant experience as a Asian American immigrant breast cancer survivor and how writing about participant experiences may affect participant's health.

DETAILED DESCRIPTION:
Primary Objective:

To determine the effects of writing therapy on QOL and perceived stress at the 6- and 12-month follow-ups.

Secondary Objective:

To discover the effects of writing therapy on stress biomarkers and perceived stress at the 3-month follow-up.

To explore the psychosocial and cultural mechanisms responsible for the benefits of writing therapy by using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 and older) diagnosed with stage 0-III cancer (or acute leukemia in remission/ chronic myeloid leukemia in chronic phase).
* Self-identified as Asian, Asian Americans, any Asian or Asian American subgroup (Chinese, Vietnamese, Indian, Korean, etc.) ethnic/cultural background
* Completed primary treatment, including surgery, chemotherapy, and/or radiation therapy, immunotherapy, or targeted therapy within the preceding 5 years.
* Comfortable reading in English or in Chinese.

Exclusion Criteria:

- Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Time Frame: through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org